CLINICAL TRIAL: NCT05383131
Title: A Single Center, Open Label Study to Evaluate Drug-drug Interactions Between HEC585 and Pirfenidone or Nintedanib in Healthy Volunteers
Brief Title: To Evaluate Drug-drug Interactions Between HEC585 and Pirfenidone or Nintedanib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HEC585-P-04 / CRC-C2032
Record Dates: First submitted 2022-05-12; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HEC585 and Pirfenidone (Experimental): period 1 - Pirfenidone X mg, TID; period 2 - HEC585 X mg, QD; period 3 - Pirfenidone X mg, TID + HEC585 X mg, QD.
  Interventions: Drug: HEC585; Drug: Pirfenidone
- HEC585 and Nintedanib (Experimental): period 1 - Nintedanib X mg, BID; period 2 - HEC585 X mg, QD; period 3 - Nintedanib X mg, BID + HEC585 X mg, QD.
  Interventions: Drug: HEC585; Drug: Nintedanib

INTERVENTIONS:
Drug: HEC585 — Mulltiple doses of HEC585 for up to 10 days
Drug: Pirfenidone — Mulltiple doses of Pirfenidone for up to 3 days
  Arms: HEC585 and Pirfenidone
Drug: Nintedanib — Mulltiple doses of Nintedanib for up to 7 days
  Arms: HEC585 and Nintedanib

SUMMARY:
An open label study to evaluate drug-drug interactions between HEC585 and Pirfenidone or Nintedanib in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

- Subjects who are willing and are able to provide a written informed consent to participate in the study.

Without Plann for pregnancy or pregnant within 3 months after enrollment throughout the trial.

Subjects aged between 18 and 45 (both inclusive) years old. Healthy volunteers has a body weight ≥50 kg (for male) or ≥ 45kg (for female in the first part of the trial) and body mass index ≥19 and ≤28 kg/m2 at screening.

Subjects, who are healthy, as having no clinically significant abnormalities in vital signs, physical examination, clinical laboratory test results, Chest X-ray and 12-lead electrocardiogram.

Exclusion Criteria:

* Subjects with a positive serology for HIV antibodies, HBsAg, HCV antibodies and/or TP antibodies at screening.

Subjects suffering from gastrointestinal diseases that can interfere with absorption or metabolism of drugs within 6 months before screening; and/or with history of central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, immune system, reproductive system; and/or thyroid disease or previous thyroid surgery, malignant tumor, metabolic disorder or others medical conditions that are not suitable for clinical trial participation.

Patients with photosensitivity and/or other skin diseases. Bleeding or thrombosis risk. Allergic. Use of any prescription or non-prescription medications within 14 days prior to initial dosing，Use of any medications known to inhibit or induce cytochrome P enzyme drug metabolism within 28 days prior to initial dosing.

Consume foods or beverages containing caffeine, xanthine, alcohol, and grapefruit within 48 hours prior to initial dosing.

Positive results from urine drug screen test. History of alcoholism or drink regularly within 3 months prior to the study. Positive for urine cotinine or smoked within 1 month before administration of study drug in the first part，regular smoking of more than 10 cigarettes per day within 3 months before administration of study drug in the second part.

Donate blood or lose blood 400 mL or more within 1 month prior to initial dosing.

Subjects who plan to receive or have had organ transplants. Females who are lactating/breastfeeding, or positive result from pregnancy test for women of child-bearing potential.

Subjects who participated in another clinical trial and have taken other study drugs within 3 months prior to initial dosing.

Any other condition with in the opinion of the investigator would render the patient unsuitable for inclusion in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Cmax of HEC585 and Pirfenidone | 0~96 hour
AUC of HEC585 and Pirfenidone | 0~96 hour
Cmax of HEC585 and Nintedanib | 0~96 hour
AUC of HEC585 and Nintedanib | 0~96 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No